CLINICAL TRIAL: NCT00847717
Title: Randomized Controlled Trial of IIb Preserving Neck Dissection VS Neck Dissections Involving IIb Removal (Selective/Functional) in Patients With N0 Neck With Oral Cavity Malignancies
Brief Title: Trial of IIb Preserving Neck Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Surgical Oncology, Banaras Hindu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SND_01
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Oral Cancer
Keywords: Oral; cancer; surgery; neck dissection; spinal accessory nerve
MeSH Terms: conditions — Mouth Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IIb preserving neck dissection
  Interventions: Procedure: Selective neck dissection
- 2 (Other): Conventional neck dissection
  Interventions: Procedure: Conventional Neck dissection

INTERVENTIONS:
Procedure: Selective neck dissection — Level IIb preserving neck dissection
  Arms: 1
Procedure: Conventional Neck dissection — Conventional neck dissection (MRND type III or Supraomohyoid)
  Arms: 2

SUMMARY:
The treatment of clinically N0 neck in malignancies of oral cavity is controversial. The options include the policy of "wait and watch"(close observation and follow-up), elective irradiation of the neck, elective surgery of the neck (neck dissection).

In elective neck dissections, the procedures commonly performed are modified radical neck dissection-III (functional neck dissection) and selective (supraomohyoid) neck dissection depending on the site of the primary lesion within the oral cavity. There are no trials of IIb preserving neck dissection in cancers of the oral cavity.

DETAILED DESCRIPTION:
Surgery of the cervical lymphatic system has evolved a lot since the introduction of classical radical neck dissection by Crile in 1906, which was later established by Martin (1945). It includes the removal of cervical lymphatic levels I-V along with removal of non-lymphatic structures namely submandibular gland, tail of parotid, omohyoid muscle, cervical plexus of nerves, spinal accessory nerve, internal jugular vein and sternocleidomastoid muscle. The main morbidity of the radical neck dissection was the trapezius muscle dysfunction with shoulder drop, resulting in pain and shoulder dysfunction. The other morbidities of radical neck dissection were cosmetic deformity of neck, painful neuromas, increased facial swelling, numbness of neck and ear.

In the last three decades, many modifications of the classical radical neck dissection (modified radical neck dissections), had been described and are increasingly applied. The main modifications have been the preservation of one or more of the non-lymphatic structures that were removed in classical radical neck dissection mainly the spinal accessory nerve, internal jugular vein, sternocleidomastoid muscle (Bocca and Pignataro, 1967). The reasons for developing these modifications were functional and cosmetic, while preserving the oncological safety of the procedure.

Much later in 1980s, the concept of selective neck dissection, for which Lindberg (1972) and Skolnik (1976) laid down important basis, was introduced. In selective neck dissections only those groups of lymph nodes are removed, which, depending upon the location of the primary tumour, are most likely to contain metastasis (Shah, 1990).

The first selective neck dissection introduced was the supraomohyoid neck dissection, which includes the removal of lymph node levels I-III, while preserving the non-lymphatic structures as functional neck dissection. Medina and Byers in a prospective study have demonstrated the utility of this supraomohyoid neck dissection in patients with clinically negative neck nodes (N0) with malignancies of oral cavity.

The posterolateral neck dissection removes lymph node levels II-V as well as retroauricular and suboccipital nodes, which is used primarily for treatment of tumours of scalp and post auricular skin.

The lateral neck dissection, which includes removal of lymph node levels II-IV, is done for tumours of larynx or hypopharynx with N0 neck.

The anterior compartment neck dissection includes removal of only lymph node level VI which is done in thyroid malignancies when there is no evidence of lateral lymphadenopathy, and is combined with lateral neck dissection(anterolateral) if there are lymphnodes involved.

Recently the concept of superselective neck dissections has been introduced. It is less radical than selective neck dissections, removing lesser number of at-risk lymph nodal groups.

H Coskun (2004) found IIb preserving superselective neck dissection as oncologically safe procedure in N0 laryngeal cancer, with more functional preservation of trapezius muscle and hence negligible shoulder disability. In this study, it was found that even in selective neck dissection, some degree of spinal accessory nerve dysfunction and shoulder disability occurs as a result of retraction of the nerve during the clearance of the lymph nodes posterior and superior to the nerve (IIb). If these lymph nodes were not removed and left in place, there would be no stretching of spinal accessory nerve during the neck dissection and shoulder disability could be avoided

ELIGIBILITY:
Inclusion Criteria:

* Patients >18yrs of age.
* histologically proven squamous cell carcinoma
* clinical and radiological N0 neck

Exclusion Criteria:

* Pregnant and lactating women

  * Patients with synchronous primaries
* H/o previous malignancy except BCC
* Previous surgeries on neck

  * Post radiotherapy recurrence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Spinal accessary nerve function | 2 years

SECONDARY OUTCOMES:
neck Node failure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, MS, Principal Investigator — Banaras Hindu University
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

REFERENCES:
- [Background] Coskun HH, Erisen L, Basut O. Selective neck dissection for clinically N0 neck in laryngeal cancer: is dissection of level IIb necessary? Otolaryngol Head Neck Surg. 2004 Nov;131(5):655-9. doi: 10.1016/j.otohns.2004.04.014. PMID 15523444
- [Background] Robbins KT, Doweck I, Samant S, Vieira F. Effectiveness of superselective and selective neck dissection for advanced nodal metastases after chemoradiation. Arch Otolaryngol Head Neck Surg. 2005 Nov;131(11):965-9. doi: 10.1001/archotol.131.11.965. PMID 16301367
- [Background] Orhan KS, Demirel T, Baslo B, Orhan EK, Yucel EA, Guldiken Y, Deger K. Spinal accessory nerve function after neck dissections. J Laryngol Otol. 2007 Jan;121(1):44-8. doi: 10.1017/S0022215106002052. Epub 2006 Jul 3. PMID 17040583
- [Background] van Wilgen CP, Dijkstra PU, Nauta JM, Vermey A, Roodenburg JL. Shoulder pain and disability in daily life, following supraomohyoid neck dissection: a pilot study. J Craniomaxillofac Surg. 2003 Jun;31(3):183-6. doi: 10.1016/s1010-5182(03)00030-1. PMID 12818606
- [Background] Taylor RJ, Chepeha JC, Teknos TN, Bradford CR, Sharma PK, Terrell JE, Hogikyan ND, Wolf GT, Chepeha DB. Development and validation of the neck dissection impairment index: a quality of life measure. Arch Otolaryngol Head Neck Surg. 2002 Jan;128(1):44-9. doi: 10.1001/archotol.128.1.44. PMID 11784253
- [Derived] Pandey M, Karthikeyan S, Joshi D, Kumar M, Shukla M. Results of a randomized controlled trial of level IIb preserving neck dissection in clinically node-negative squamous carcinoma of the oral cavity. World J Surg Oncol. 2018 Nov 8;16(1):219. doi: 10.1186/s12957-018-1518-z. PMID 30409212